CLINICAL TRIAL: NCT06368752
Title: GA-18: The Role of Endogenous GIP in Glycosis Metabolism During Fasting
Brief Title: The Role of Endogenous GIP in Glycosis Metabolism During Fasting
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Frederikke Koefoed-Hansen (Other)
Responsible Party: Sponsor-Investigator, Frederikke Koefoed-Hansen, Research Student, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-22063621
Record Dates: First submitted 2023-07-30; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — gastric inhibitory polypeptide (3-30)-amide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The trial is a randomized, double-blind, crossover study. We give intravenous infusion of GIP[3-30]NH2, and thus describe the effects of GIP by comparing with what happens during a saline infusion (placebo).
Who Masked: Participant, Investigator
Masking Description: The infusion is mixed by an external coordinator. Neither the investigator or the participants knows whether is the GIP[3-30]NH2 infusion or saline infusion that is being given. Which infusion that is given on each trial day is randomized for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIP[3-30]NH2 infusion (Experimental): GIP[3-30]NH2 intravenous infusion (800 pmol/kg/min)
  Interventions: Biological: GIP[3-30]NH2
- Saline infusion (Placebo Comparator): Saline intravenous infusion (0,5 % human serum albumin)
  Interventions: Other: Saline

INTERVENTIONS:
Biological: GIP[3-30]NH2 — GIP[3-30]NH2 is the naturally occurring shorter (truncated) variant of GIP[1-42]. GIP[3-30]NH2 also stimulates the GIP receptor and therefore acts like a GIP receptorantagonist
  Arms: GIP[3-30]NH2 infusion
Other: Saline — Sodium chlorid with 0,5% human serum albumin.
  Arms: Saline infusion

SUMMARY:
This research project aims to investigate the role of endogenous GIP during fasting. With the infusion of a GIP receptor antagonist (GIP[3-30]NH2), is it possible to selectively remove the effect of endogenous GIP, and thus describe its effects by comparing it with what happens during a saline infusion.

DETAILED DESCRIPTION:
This research project investigates the effects endogenous GIP has in the body of healthy, overweight people. Two trial days will be held. The participant will receive intravenous infusion of either GIP[3-30]NH2 (800 pmol/kg/min) or placebo (saline) in a randomized order. After 20 minutes, GIP[3-30]NH2 is expected to have maximum effect. On time of 180 minutes, an ad libitum meal is served, which is consumed during continued infusion. When the participant is comfortably full, the infusion is turned off and the trial day ends. During the day, the participant assesses and notes on standardized VAS schedules current appetite, satiety, nausea, fatigue, malaise and thirst. Blood pressure and heart rate are measured every 30 minutes throughout the trial day and blood samples are taken. In total, there will be drawn ten blood samples between intervals of 15 to 30 min. Three times along the way, the activity in the brown adipose tissue is measured with a thermal camera (temperature measurements over the skin on the chest) and the resting metabolic rate is determined with indirect calorimetry (inhaled and exhaled air is captured by breathing under a large plastic bell).

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* BMI > 30 kg/m2
* Body fat percentage > 25 % for men og > 35 % for women

Exclusion Criteria:

* Type 1 diabetes and/or type 2 diabetes diagnosis
* Other chronic condition
* Treatment with medications or supplements that cannot be paused for 12 hours
* > 14 units of alcohol weekly or drug abuse
* Circulating liver enzymes (alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT)) ≥ 2 × normal value
* Renal impairment (eGFR < 90 or creatinine level above the reference range)
* Uncontrolled high resting blood pressure (above 140/90 mmHg)
* Low blood percentage (hemoglobin < reference range (different for women and men))
* Special diet or planned weight change within the trial period
* Any disease/condition that investigators believe will interfere with study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma glucagon concentrations | Four hours
  Measured in mmol/L. The primary endpoint is plasma glucagon concentrations during GIP[3-30]NH2 infusion compared to placebo.Area under the curve (AUC) for plasma glucagon (AUCglucagon) is quantified both as absolute and in baseline-subtracted values (bsAUCglucagon) and the effect of the GIP receptor antagonist will be calculated as a percentage reduction of bsAUC glucagon relative to bsAUC glucagon during the placebo infusion.

SECONDARY OUTCOMES:
Plasma levels of C-peptide | Four hours
  Measured in mmol/L
Plasma levels of insulin | Four hours
  Measured in mmol/L
Resting metabolic rate | 15 minutes
  Measured in resting energy expenditure (REE) and respiratory quotient (RQ)
Activity in brown adipose tissue | 10 minutes
  Measured by thermal camera
Appetite | 30 minutes
  Measured in kilogram food intake
Blood pressure | Pre-intervention at time -30 and -20 min. During infusion at time 0 min, 30 min, 60 min, 90 min, 120 min, 160 min and 180 min.
  mmHg
Puls | Pre-intervention at time -30 and -20 minutes. During infusion at time 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 160 minutes, and 180 minutes
  Beats pr. minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The results of this project or sub-elements of the project will be compiled into one or more manuscripts for publication in one or more international scientific high impact journals. All results, both inconclusive, negative and positive trial results, will be published as soon as possible. All trial participants will be informed in writing of the results after the end of the trial.
Supporting Information: CSR
Time Frame: December 31st. 2025

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT06368752/Prot_SAP_000.pdf